CLINICAL TRIAL: NCT05623163
Title: Evaluation of Health Improvement in Obese Patients With Obesity-related Comorbidities Followed by EndoZip Procedure
Acronym: CL00010
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nitinotes Surgical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CL00010
Record Dates: First submitted 2022-11-06; First posted 2022-11-21 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EndoZip System (Experimental): The Nitinotes EndoZip system is designed to allow for the creation of multiple internal gastric segmentation (up to 5) in the stomach by using an endoscopic approach. The system allows the forming of wall-to-wall longitudinal attachments of the anterior and posterior stomach walls, creating multiple strictures within.
  Creation of this segmentation may significantly reduce gastric volume, may affect gastric motility and consequently, reduce weight.
  Interventions: Device: EndoZip System

INTERVENTIONS:
Device: EndoZip System — The Nitinotes EndoZip system is designed to allow for the creation of multiple internal gastric segmentation (up to 5 sutures) in the stomach by using an endoscopic approach. The system allows the forming of wall-to-wall longitudinal attachments of the anterior and posterior stomach walls, creating multiple strictures within.
  Creation of this segmentation may significantly reduce gastric volume, may affect gastric motility and consequently, reduce weight.

SUMMARY:
multicenter, prospective, single arm study will include up to 45 patients, (up to 30 patients per site), aimed at evaluating the performance of the EndoZip System in obese patients with type 2 diabetes and / or hypertension who failed to reduce weight with non-surgical weight-loss methods.

Patients will be enrolled in 2 clinical sites in Europe. Patients who meet the eligibility criteria is expected to come the clinic for at least 10 visits.

DETAILED DESCRIPTION:
study will include up to 45 (up to 30 patients per site), ages of 21 -75 of obese patients (BMI 30-40 kg/m²) who failed to reduce weight with non-surgical weight-loss methods.

At least 50% of the population included in the study diagnosed with Type 2 diabetes (T2D), and with HbA1c < 9 at least 6 months prior to study enrollment, excluding Insulin-dependent and / or At least 50% of the population included in the study diagnosed with hypertension, treating with 2 or more antihypertensive medications and are well control at least 6 months prior to study enrollment.

The duration for each participant will be 12 months and will include the following follow up visits and procedures:

* Office visits: screening, procedure day, 1 week, and 1, 2, 4, 6, 8, 10, and 12 month(s)
* Remote follow up (by Phone): 3, 5, 7, 9, and 11 month(s)
* Endoscopy: procedure day and 2 months
* Electrocardiogram (ECG) test: Screening and procedure day
* FibroScan test: Screening, 6 and 12 months
* 24- hours Home Ambulatory Blood Pressure Monitor (ABPM), only for patients diagnosed with hypertension: Screening, 6 and 12 months
* Laboratory tests including: (1) Hematology blood tests, (2) Biochemistry blood tests for: sugar Metabolism, liver, proteins, and lipid (3) Urinalysis (Dipstick) tests: Screening, 6 and 12 months.
* Physical examination (include at minimum examination of: GI, Cardiopulmonary, Hepatobiliary and extremities systems) - Screening and procedure day.
* Vital signs (blood pressure and heart rate - supine, pulse, body temperature, respiratory rate (RR) and SpO2): Screening, procedure day, 1 week, 1, 2, 4, 6, 8, 10 and 12 months
* BMI and Waist circumference: Screening, procedure day, 1 week, 1, 2, 4, 6, 8, 10 and 12 months
* Meeting with dietitians / lifestyle modifications counseling: at all follow up office and remote visits:

  * Office visit: Screening, procedure day, 1 week, 1, 2, 4, 6, 8, 10 and 12 months
  * Remote follows up (phone calls) at months 3,5,7,9, and 11.
* IWQOL-Lite: Screening, 2, 6 and 12 months
* PHQ-9: Screening
* Pregnancy test (only for the relevant population): Procedure day

The patient will required to follow a specific diet and to have a physical activity during the study period ( 12 month).

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-75
2. BMI ≥ 27 and ≤40 kg/m².
3. Willingness to comply with the substantial behavioral modifications and dietary restrictions as required by the procedure.
4. Patients with history of failure with non-surgical weight-loss methods.
5. Willingness to follow protocol requirements, including signed informed consent, routine follow-up schedule, completing laboratory tests, completing IWQOL questionnaire and completing the medically supervised diet and behavior modification program.
6. Ability to give informed consent.
7. Women of childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods.
8. At least 50% of the population included in the study diagnosed with Type 2 diabetes (T2D), and with HbA1c < 9 at least 6 months prior to study enrollment, excluding Insulin-dependent.
9. At least 50% of the population included in the study diagnosed with hypertension, treating with 2 or more antihypertensive medications and are well control at least 6 months prior to study enrollment.

Exclusion Criteria:

1. Prior surgery of any kind on the gastrointestinal tract (except uncomplicated cholecystectomy or appendectomy).
2. Patients with history of small bowel or colonic obstruction, and/or adhesive peritonitis and/or abdominal adhesions.
3. Patients with any inflammatory disease
4. Patients with history of cancer in the gastrointestinal tract.
5. Potential upper gastrointestinal bleeding conditions such as a history of angioectasias.
6. A known gastric mass or gastric polyps > 1 cm in size.
7. Patients with TG >500 or LDL >190
8. Patients with BP >180 / 110
9. A known hiatal hernia > 4cm of axial displacement of the z-line above the diaphragm or severe or intractable gastro-esophageal reflux symptoms while on maximal medical therapy.
10. A structural abnormality in the esophagus or pharynx such as a stricture or diverticulum that could impede passage of the endoscope.
11. Patient with motility disorders of the GI tract or intractable constipation
12. Patients with known coagulation disorder (INR >1.5) or on anticoagulation therapy.
13. Type 1 diabetes or Type 2 diabetes with a HgbA1c >9 and/or injectable medications or likely requiring insulin treatment in the following 12 months.
14. Patients with any serious health condition unrelated to their weight that would increase the risk of endoscopy
15. Patients with chronic abdominal pain
16. Patients with hepatic insufficiency or cirrhosis (CAB>290 Db/m or Fibrosis score >10 kPa)
17. Patients with viral and / or autoimmune hepatitis
18. Presence of any other form of chronic liver disease
19. Recent (within 12 months) or concomitant use of agents known to cause hepatic steatosis (long-term systemic corticosteroids [>10 days], amiodarone, methotrexate, tamoxifen, tetracycline, high dose oestrogens, valproic acid)
20. Any contraindication to liver biopsy
21. Recent (within 3 months) change in dose/regimen or introduction of Vitamin E (at a dose of ≥400 IU/day), betaine, s-adenosyl methionine, ursodeoxycholic acid, silymarin or pentoxifylline
22. Patients that used an intragastric device for weight loss
23. Patients with psychological health questionnaire-9 (PHQ-9) score of 10 or higher.
24. Patients receiving daily prescribed treatment with high dose aspirin (> 100mg daily), anti-inflammatory agents, anticoagulants or other gastric irritants or on low dose aspirin and cannot come of medication for a total of 10 days peri procedure.
25. Patients with history or current abuse of drugs or alcohol
26. Patients who are unable or unwilling to take prescribed Proton Pump Inhibitor (PPI) medication
27. Patients who are pregnant or breast-feeding.
28. Patients who are taking medications that cause weight loss within the last 6 months
29. Patients with Severe cardiopulmonary disease or other serious organic disease which might include known history of coronary artery disease, Myocardial infarction within the past 12 months and / or poorly-controlled hypertension
30. Patients are currently on medications that are known to affect gastric emptying, such as anti-seizure or anti-arrhythmic medications and / or poorly-controlled Glycemia
31. Patients who are taking corticosteroids, immunosuppressants, or narcotics and cannot come of medication for the study period.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Percent of total body weight loss (%TBWL) after 12 months. | 12 months
  percent of TBWL from baseline (prior to EndoZip procedure) and 12 month post EndoZip
Percent of patients with a reduction in %TBWL of at least 10% at 12 months | 12 months
  Percentage of patients with a reduction in %TBWL of at least 10% at 12 months
safety evaluation- Rate of adverse events | 12 months
  The cumulative incidence of adverse events observed during the procedure and throughout the follow-up period, will be presented in tabular format. A detailed list of all adverse events will be presented. The adverse event rate will be compiled with respect to seriousness, severity, expectedness and relationship to procedure and device.

CONTACTS AND LOCATIONS:
Overall Officials: Ravit Peled, Study Director — NiTiNotes Ltd
Locations (2):
- IKEM MC, Prague, Praha 4, Czechia
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No